CLINICAL TRIAL: NCT02642952
Title: Impact of Aortic Grafts After Open and Endovascular Repair in Central Hemodynamics and Arterial Stiffness Measured by Non-invasive Methods in Patients With Abdominal Aortic Aneurysms.
Brief Title: Impact of Grafts and Endografts for Abdominal Aneurysms on Arterial Stiffness.
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Andrés Reyes Valdivia, Vascular Surgery Consultant. MD, FEBVS, Hospital Universitario Ramon y Cajal
Other Study IDs: IMPACT001
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-08

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: arterial stiffness, central hemodynamics
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Open-graft group: Patients treated for abdominal aortic aneurysm with open graft will be measured for central hemodynamics and arterial stiffness by non-invasive methods.
  Interventions: Other: non-invasive methods
- Endograft group: Patients treated for abdominal aortic aneurysm with endograft will be measured for central hemodynamics and arterial stiffness by non-invasive methods.
  Interventions: Other: non-invasive methods

INTERVENTIONS:
Other: non-invasive methods — To measure central hemodynamics and arterial stiffness by non-invasive methods using SphygmocoR (Atcor Medical, Sydney, Australia) before and after the procedure.

SUMMARY:
The purpose of this study is to evaluate by non-invasive methods the change in central hemodynamics and arterial stiffness produced by grafts and endografts after abdominal aortic aneurysm repair.

Our main goal is to measure the changes in:

Augmentation index, central blood pressure, pulse wave analysis, pulse wave velocity.

DETAILED DESCRIPTION:
The measures will be done before the procedure and after them.

We will use the device called: SphygmocoR (Atcor Medical, Sydney, Australia).

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of abdominal aortic aneurysm requiring repair (open or endovascular) based on guidelines criteria for management.

Exclusion Criteria:

* Patients who don´t want to enter in the study.
* Patients who don´t want to sign the informed consent.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consecutive treated for abdominal aortic aneurysm. The election of treatment is selected based on morphology and health status.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Reyes, Consultant, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Vascular Surgery Department, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paraskevas KI, Bessias N, Psathas C, Akridas K, Dragios T, Nikitas G, Andrikopoulos V, Mikhailidis DP, Kyriakides ZS. Evaluation of aortic stiffness (aortic pulse-wave velocity) before and after elective abdominal aortic aneurysm repair procedures: a pilot study. Open Cardiovasc Med J. 2009 Dec 9;3:173-5. doi: 10.2174/1874192400903010173. PMID 20054420
- [Background] Kadoglou NP, Moulakakis KG, Papadakis I, Ikonomidis I, Alepaki M, Lekakis J, Liapis CD. Changes in aortic pulse wave velocity of patients undergoing endovascular repair of abdominal aortic aneurysms. J Endovasc Ther. 2012 Oct;19(5):661-6. doi: 10.1583/JEVT-12-3916MR.1. PMID 23046333
- [Background] Kadoglou NP, Moulakakis KG, Papadakis I, Ikonomidis I, Alepaki M, Spathis A, Karakitsos P, Lekakis J, Liapis CD. Differential effects of stent-graft fabrics on arterial stiffness in patients undergoing endovascular aneurysm repair. J Endovasc Ther. 2014 Dec;21(6):850-8. doi: 10.1583/14-4772MR.1. PMID 25453890
- [Background] Lantelme P, Dzudie A, Milon H, Bricca G, Legedz L, Chevalier JM, Feugier P. Effect of abdominal aortic grafts on aortic stiffness and central hemodynamics. J Hypertens. 2009 Jun;27(6):1268-76. doi: 10.1097/HJH.0b013e3283299b22. PMID 19342960
- [Derived] Valdivia AR, Fuente MF, Santos AD, Urena MG, Lozano AR, Guaita JO, Zuniga CG, Donas K, Ruiz JS. Impact of the Aortic Graft on Arterial Stiffness and Inflammatory Biomarkers after Endovascular Aortic Repair or Open Surgical Repair in Abdominal Aortic Aneurysm Disease. Ann Vasc Surg. 2019 Aug;59:84-90. doi: 10.1016/j.avsg.2018.12.092. Epub 2019 Feb 23. PMID 30802592

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-graft Group | Endograft Group
Started | 21 | 30
Completed | 19 | 25
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-graft Group | Endograft Group | Total
Number analyzed (Participants) | 19 | 25 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (6.9) | 77.4 (7.2) | 74.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 18 | 23 | 41
Diameter AAA (mm) [Mean (Standard Deviation); unit: mm] | 54 (5.1) | 63.2 (12.1) | 59.3 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Aix@75
Description: Augmentation Index corrected to 75 bpm
Time Frame: Before surgery
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open-graft Group | Endograft Group
Number analyzed (Participants) | 19 | 25
percentage | 31.8 (8.9) | 32.5 (7.7)

2. Primary Outcome: AIx@75
Description: Augmentation Index corrected to 75 bpm
Time Frame: 2 months after Surgery
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open-graft Group | Endograft Group
Number analyzed (Participants) | 19 | 25
percentage | 29.3 (7.5) | 28.4 (9.2)

3. Secondary Outcome: Central Blood Pressure
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Open-graft Group | Endograft Group
Number analyzed (Participants) | 19 | 25
mmHg | 120.8 (17.8) | 122.7 (16.1)

4. Secondary Outcome: Carotid Radial Pulse Wave Velocity
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: cm/seg
Arm/Group | Open-graft Group | Endograft Group
Number analyzed (Participants) | 19 | 25
cm/seg | 7.99 (1.44) | 8.41 (1.6)

5. Secondary Outcome: Carotid Radial Pulse Wave Velocity
Time Frame: 2 months after surgery
Measure: Mean (Standard Deviation); unit: cm/seg
Arm/Group | Open-graft Group | Endograft Group
Number analyzed (Participants) | 19 | 25
cm/seg | 8.01 (1.4) | 8.17 (0.9)

ADVERSE EVENTS:
Arm/Group | Open-graft Group | Endograft Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/25
Other Adverse Events (participants affected / at risk) | 0/19 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes